CLINICAL TRIAL: NCT01740973
Title: Risk of Umbilical Trocar-site Hernia After SILC Versus Conventional Laparoscopic Cholecystectomy
Brief Title: Risk of Umbilical Trocar-site Hernia After SILC Cholecystectomy Versus Conventional Cholecystectomy
Acronym: UMBI-SILS
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, M. D., Hvidovre University Hospital
Other Study IDs: UMBI-SILS-123
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Cholecystolithiasis; Incisional Hernia
Keywords: SILC; lap. cholecystectomy; trocar-site hernia
MeSH Terms: conditions — Cholecystolithiasis; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SILC cholecystectomy: No intervention. 239 SILC having a prospective questionnaire and clinical follow-up, if the patient suspects an umbilical hernia.
- and conventional lap. cholecystectomy: no intervention.Patients are also mailed a prospective questionnaire and clinical follow-up, if the patient suspects an umbilical hernia.

SUMMARY:
Background Laparoscopic cholecystectomy is a very common procedure. Postoperative pain, especially around the umbilical port is dominating the first postoperative week. Single Incision Laparoscopic cholecystectomy (SILC) has been proposed to diminish postoperative incisional pain and improve cosmetic results, but results are not convincing and the risk of formation of an umbilical trocar-site hernia is not properly investigated.

This study aimed to investigate the risk of umbilical trocar-site hernia formation after SILC vs. conventional 4-port laparoscopic cholesystectomy.

Methods This is a cohort registry study with prospective questionnaire and clinical follow-up on 239 patients having a SILC from 1/1 2009 to 1/6 2011 vs. 478 mathed patients having a conventional laparoscopic cholecystectomy (consecutively from one month before and after SILC. They are matched for age, gender, date of operation, and surgeons skills (database from intraoperatively registered data). Primary endpoint is umbilical trocar-site hernia formation (operation for a umbilical hernia or clinical hernia).

The H0 hypothesis is that there is not difference between SILC and conventional.

Exclusion criteria are: death, operation for acute cholecystitis. The included patients will be sent a questionnaire asking for operation for a hernia in the area, suspicion of a hernia, and perioperative data that we do not have in the database. Futhermore those patients who suspect a hernia will be invited to aclinical exam by a medic to state the diagnosis. Furthermore we patients are asked to report if they have chronic pain and/or discomfort.

ELIGIBILITY:
Inclusion Criteria:

* SILC 1/1-2009-1/6-2011 and matched controls consecutively from the cholecystectomy-database having a lap. chol. one month before and one month after the SILC group.

Exclusion Criteria:

* death in the follow-up time
* an abdominal operation before la.chol/SILC with midline incision
* an abdominal operation after la.chol/SILC with midline incision
* primary operation for acute cholecystitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient having a SILC in Denmark from 1/1-2009-1/6-2011 and matched conventional lap. cholecystectomies. Matched in gender, age, surgeons ecxperience
Sampling Method: Non-Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Umbilical trocar-site hernia formation | participants will be followed for expected average of 3 years
  Operation for an umbilical trocar-site hernia or clinical trocar-site hernia formation

SECONDARY OUTCOMES:
chronic pain and discomfort | participants will be followed for expected average of 3 years
  The degree of long-term chronic pain and discomfort after cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Mette w Christoffersen, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark